CLINICAL TRIAL: NCT05423912
Title: Keeping on Course: A Communication-Focused Psychoeducation Program for Dyads Coping With Mild Cognitive Impairment
Brief Title: Keeping on Course: A Communication-Focused Psychoeducational Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Emory University (Other)
Collaborators: National Institute on Aging (NIA) (NIH); Emory Roybal Center for Dementia Caregiving Mastery (Unknown)
Responsible Party: Principal Investigator, Kenneth Hepburn, Professor, Emory University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: STUDY00003645; P30AG064200 (NIH)
Record Dates: First submitted 2022-06-01; First posted 2022-06-21 (Actual); Last update posted 2026-01-27 (Actual); Status verified 2026-01

CONDITIONS: Mild Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Intervention Model Description: Participants are 24 dyads of persons with MCI and their care partners who experience the same intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Keeping on Course Program for Persons with Mild Cognitive Impairment (MCI) (Experimental): Persons with MCI participating in the Keeping on Course program.
  Interventions: Behavioral: Keeping on Course Program
- Keeping on Course Program for Care Partners of MCI Participants (Experimental): Care partners participating in the Keeping on Course program with the MCI participant they care for.
  Interventions: Behavioral: Keeping on Course Program

INTERVENTIONS:
Behavioral: Keeping on Course Program — MCI dyads engaging in the testing aim of the Keeping on Course Program take part in group meetings lasting 90 to 120 minutes over the course of 6 virtual meetings. Participants are asked to take part in structured quantitative interviews at baseline and 4 and 8 weeks post-intervention. A subsample of participants will be invited to take part in a virtual, semi-structured 30-60 minute qualitative interview focused on their experiences in and perceptions of the intervention.

SUMMARY:
The goal of Keeping on Course is to develop and test a psychoeducation program to provide dyads facing mild cognitive impairment (MCI) with communication skills and strategies that will establish or restore a sense of agency as they cope with MCI.

DETAILED DESCRIPTION:
Up to 21% of older adults exhibit symptoms of mild cognitive impairment (MCI), a term used to describe a compilation of cognitive and behavioral symptoms that approach but don't meet the threshold for a dementia diagnosis. Noticeably characterized by losses in executive function and memory that can affect critical life domains like employment, housing, health care, and finances, it is also a life condition of considerable indeterminacy both for the person living with the condition and for care partners. While many individuals experience worsened symptoms leading to an Alzheimer's disease (AD) diagnosis within five years, MCI can be caused by a variety of disease processes making disease trajectory and prognosis vague and uncertain.

For most diagnosed with MCI, the experience is shared with another, typically a spouse or partner. In many cases, other members of the family, including fictive kin, are part of the team providing care and support - not only to the person living with MCI but to the principal caregiver, as well. For the dyad and both parties in an MCI couple individually, the period following an MCI diagnosis is often one of extended emotional turbulence and ambiguity. Care partner dyads coping with MCI face changes in role identity resulting in significant consequences for relationships, and the turbulence extends beyond the dyad to the larger extended family. It is unclear what the future might hold or how pervasively established patterns of living will be altered. The foundations of shared expectations and of trustworthy methods of planning, communication, and decision-making are disrupted in unpredictable ways. Emotional adjustment to MCI, unique for each dyad, has implications for subsequent family coping, psychological stress, physical fatigue, social isolation, decision-making, financial well-being, and more.

While MCI psychoeducation programs exist, they almost always target the person with MCI and not the patient-care partner dyad. Communication patterns between patients and care partners in oncology and HIV/AIDS settings are shown to influence the coping and care outcomes of dyads. With similar communication issues noted in MCI dyads, the goal of this pilot project is to develop and test the feasibility and preliminary efficacy and evaluate acceptability of a group program, Keeping on Course, to provide couples facing MCI with communication skills and interpersonal strategies that will establish or restore a sense of agency and emotional well-being as they navigate this period of transition and uncertainty.

This study uses a one-arm, pre/post design to assess the acceptability, feasibility, and preliminary efficacy in 4 cohorts of 6 MCI dyads each (for a total of 48 individuals) to take part in a trial of the Keeping on Course program. Participants meet in virtual intervention group meetings over the course of 6 consecutive weeks. Participants are asked to take part in structured quantitative interviews prior to the intervention and then 4 and 8 weeks post-intervention.

ELIGIBILITY:
Inclusion Criteria:

* Either a person with MCI, defined as a score of 23-27 on the Mini-Mental State Examination (MMSE) or a score of 19-25 on the Montreal Cognitive Assessment (MoCA), or an MCI care partner
* Can read, speak, and understand English
* Have internet connectivity and a separate zoom-enabled device for each dyad member
* Dyads must live together, as this will provide sufficient opportunity for intervention homework and communication practice activities

Exclusion Criteria:

* Individuals who are not yet adults (infants, children, teenagers)
* Pregnant women
* Prisoners
* Individuals who are not able to clearly understand and speak English
* Those living with MCI will need to successfully complete a capacity to consent survey to be included in the study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2023-02-08 (Actual); Primary Completion 2025-12-08 (Actual); Study Completion 2025-12-08 (Actual)

PRIMARY OUTCOMES:
Acceptability of Intervention Measure (AIM) Score | 4 weeks post-program, 8 weeks post-program
  Acceptability, appropriateness, and feasibility of the Keeping on Course program are assessed with three items from the Acceptability of Intervention Measure (AIM). Items are scored on a 5-point scale where "completely disagree" = 1 and "completely agree" = 5. The total score is the average score of all items and ranges from 1 to 5. Higher scores indicate greater acceptability of the intervention.
Intervention Appropriateness Measure (IAM) Score | 4 weeks post-program, 8 weeks post-program
  Appropriateness of the Keeping on Course program is assessed with three items from the Intervention Appropriateness Measure (IAM). Items are scored on a 5-point scale where "completely disagree" = 1 and "completely agree" = 5. The total score is the average score of all items and ranges from 1 to 5. Higher scores indicate greater appropriateness of the intervention.
Awareness, Courage, and Responsiveness Scale Score | 4 weeks post-program, 8 weeks post-program
  The Awareness, Courage, and Responsiveness Scale asks 24 questions to measure awareness of others, self-awareness, courage, and responsiveness towards others. Responses to survey items are given on a 7-point scale where "never true" = 1 and "always true" = 7. The total score ranges from 24 to 168. Higher scores indicate greater expression of interpersonal dynamics of being aware, courageous in uncomfortable situations, and being responsive to the needs of others.
Feasibility of Intervention Measure (FIM) Score | 4 weeks post-program, 8 weeks post-program
  Feasibility of the Keeping on Course program is assessed with three items from the Feasibility of Intervention Measure (FIM). Items are scored on a 5-point scale where "completely disagree" = 1 and "completely agree" = 5. The total score is the average score of all items and ranges from 1 to 5. Higher scores indicate greater feasibility of the intervention.
Attendance | Up to Week 6
  Feasibility of the intervention is assessed with the number of sessions attended.
Completion of Homework Assignments | Up to Week 6
  Feasibility of the intervention is assessed with the number of homework assignments completed.
Group Participation | Up to Week 6
  Feasibility of the intervention is assessed with the number of participants engaging in group activities.
Percent of Participants Completing Surveys | Baseline, 4 weeks post-program, 8 weeks post-program
  Acceptability of measurements used to understand decision-making in dyads coping with MCI is assessed as the completion rates of each of four instruments. An instrument is considered acceptable if there is a 90% completion rate for an instrument.

SECONDARY OUTCOMES:
Perceived Stress Scale (PSS-14) Score Among Care Partners | Baseline, 4 weeks post-program, 8 weeks post-program
  The 14-item Perceived Stress Scale (PSS-14) is a measure of the degree to which situations in one's life are appraised as stressful. Care Partner participants are asked questions about their thoughts and feelings during the last month. Responses are given on a 5-point scale where "never" is scored as 0 and "very often" is scored as 4. Total scores range from 0 to 56 with higher scores indicating greater perceived stress.
Midlife Development Inventory (MIDI) Sense of Control Scale | Baseline, 4 weeks post-program, 8 weeks post-program
  The Midlife Development Inventory (MIDI) Sense of Control Scale asks respondents to assess their sense of control over their life. The 12 items are responded to on a 7-point scale where "strongly agree" = 1 and "strongly disagree" = 7. A total score is obtained by calculating the average score of all items. When calculating a total score, certain items are reversed. Total scores range from 1 to 7 with lower scores indicate greater sense of control over life.
Decision-Making Involvement Scale | Baseline, 4 weeks post-program, 8 weeks post-program
  The Decision-Making Involvement Scale is administered to participants with MCI and their care providers. The instrument assesses the agency in personal decision-making of the person living with mild cognitive impairment with 5 items. Responses to items are given on a 4-point scale where "not at all involved" = 0 and "very involved" = 3. Total scores range from 0 to 15 with higher scores indicating the participant with MCI has greater involvement with personal decision-making.
Decision-Making Involvement Measure | Baseline, 4 weeks post-program, 8 weeks post-program
  A modified version of the Decision-Making Involvement Measure is used in this study to assess participation in the discussions during the Keeping on Course program. The first five items are responded to on a 4-point scale where "none/never" = 1 and "all/always" = 4. Total scores range from 5 to 20 with higher scores indicating greater feelings of involvement in the program discussions.
Decision-Making Involvement Measure - Overall Satisfaction | Baseline, 4 weeks post-program, 8 weeks post-program
  A modified version of the Decision-Making Involvement Measure is used in this study to assess participation in the discussions during the Keeping on Course program. Item 6 asks participants how satisfied they were with the series of discussions overall. Responses are given on a 7-point scale where "not very well at all" = 0 and "very well indeed" = 6.

CONTACTS AND LOCATIONS:
Overall Officials: Kenneth Hepburn, PhD, Principal Investigator — Emory University
Locations (1):
- Emory Clinic at Executive Park, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: Yes
The de-identified dataset, including common measures of care partner self-efficacy and mastery, as well as certain demographic data, will be made available for sharing with other researchers.
Supporting Information: Study Protocol
Time Frame: Data will be made available for sharing once the main findings from this study are published.
Access Criteria: Data from this pilot study will be available to qualified researchers through a data sharing agreement that is fully consistent with NIH data sharing policies and applicable laws and regulations as well as official policies and practices established. Study data will be deposited in the Roybal Center data repository. Data will be made available to qualified researchers via an NIH-approved data sharing agreement.
  The data sharing agreement will require:
  1. a commitment only to use the data for research purposes and not to identify any individual participant;
  2. a commitment to securing the data using appropriate computer technology; and
  3. a commitment to destroy or return the data after analyses are completed.
  Analyses will be up to the discretion of the requesting researcher and restrictions outlined in the data sharing agreement.

DOCUMENTS (1):
  • Informed Consent Form (2025-01-05): https://cdn.clinicaltrials.gov/large-docs/12/NCT05423912/ICF_000.pdf